CLINICAL TRIAL: NCT05695378
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate the Efficacy and Safety of KM-819 Treatment to Slow the Progression of Multiple System Atrophy
Brief Title: Trial to Evaluate the Efficacy and Safety of KM-819 Treatment to Slow the Progression of Multiple System Atrophy (MSA)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor has decided to withdraw the study due to safety issue and re-initiate with a new clinical study
Sponsor: Kainos Medicine Inc. (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KMCP-819-K102
Record Dates: First submitted 2022-12-22; First posted 2023-01-25 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Multiple System Atrophy
Keywords: neurodegenerative disorder; Fas-associated factor 1 (FAF1); autonomic dysfunction; KM-819
MeSH Terms: conditions — Multiple System Atrophy; Neurodegenerative Diseases; Primary Dysautonomias | interventions — KM-819

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Main Study: KM-819 (Experimental): Subjects will receive 400 mg of KM-819 orally from Week 0 to Week 36.
  Interventions: Drug: KM-819
- Main Study: Placebo (Placebo Comparator): Subjects will receive visually identical placebo pills of KM-819 orally.
  Interventions: Drug: Placebo
- Ancillary Study: KM-819 (Experimental): Subjects will receive 400 mg of KM-819 orally from Week 40 to Week 76.
  Interventions: Drug: KM-819

INTERVENTIONS:
Drug: KM-819 — Subjects will receive KM-819 400 mg orally daily.
  Arms: Ancillary Study: KM-819; Main Study: KM-819
Drug: Placebo — Subjects will receive Placebo orally daily.
  Arms: Main Study: Placebo

SUMMARY:
This trial will the efficacy of KM-819 compared to placebo in subjects with MSA for slowing the progression of MSA.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled phase II trial. This trial will be performed in two part: Main study and Ancillary study.

Main Study: Following a 4-week screening period, subjects will be stratified by MSA subtype (MSA-P, -C [MSA-Parkinsonian type, MSA-cerebellar ataxia]) and randomly assigned in a 1:1 ratio either to KM-819 or Placebo groups.

During a treatment period of 36 weeks, subjects will receive pills of either KM-819 or Placebo for oral administration every day from baseline visit. Following this, there will be a safety follow-up period at Week 40.

Ancillary Study: This ancillary study will provide additional information on the continuing efficacy and safety of KM-819. Subjects in either treatment group in the main study who complete the study are eligible to participate in a follow-up, all-subjects-on-treatment (KM-819), open-label ancillary study.

All subjects in the ancillary study will receive KM-819 for additional 36 weeks regardless of their treatment allocation during the main study. During a treatment period of 36 weeks, subjects will receive pills of KM-819 for oral administration every day from visit at Weeks 40.

ELIGIBILITY:
Inclusion Criteria:

1. Must be diagnosed as probable or possible MSA, according to the second consensus criteria for diagnosis of MSA
2. Patients who are able to visit the clinic during the study period to be in the study.
3. ≥ 30 years and ≤ 80 years of age at the time of signing the Informed Consent
4. Antiparkinsonian medications should be stable for, at least, one month before enrollment.
5. Body Mass Index (BMI) range of 18.5 to 30 kg/m^2 inclusive at Screening
6. Patient agrees to use acceptable contraceptive methods during the study
7. For women, menopause, sterilization confirmed.
8. For childbearing women, older than 40, and agreed with more than 2 methods of contraception below and agreed with no desire to be pregnant during and after the study, and, agreed with maintaining medically acceptable methods of contraception during for 90 days after the study.
9. Cognitive ability for possible to make self-decision, understand and follow the instruction, to make written signature on consent form.
10. If no ability to walk, patients must be accompanied by caregiver by wheelchair on schedule.

Exclusion Criteria:

1. A diagnosis of drug induced parkinsonism by typical neuroleptic treatment or haloperidol medication.
2. Women who are pregnant or lactating
3. History of suicide attempt. Any recent suicidal ideation (a level of 4 or 5) within the last 3 months prior to Day 1, or has a positive response ('Yes') to either question 4 or 5 of the Columbia Suicide Severity Rating Scale (C-SSRS) at check-in (Day 1), or who is at significant risk to commit suicide, as judged by the Investigator using the C-SSRS at Screening.
4. Febrile illness or symptomatic viral, bacterial (including upper respiratory infection) or fungal (non-cutaneous) infection.
5. Any clinically significant abnormality following the Investigator's review of the physical examination and protocol-defined clinical laboratory tests at Screening or site check-in.
6. Patient has a mean pulse rate < 40
7. Patient has a mean corrected QT interval using Fridericia's formula (QTcF) of > 430 msec (for males) and > 450 msec (for females).
8. History of unexplained syncope, cardiac arrest, unexplained cardiac arrhythmias or torsade de pointes, structural heart disease or a family history of Long QT Syndrome.
9. Positive serology test for hepatitis B surface antigen (HBsAg), anti-hepatitis A virus (HAV), immunoglobulin M (IgM), anti-hepatitis C virus (HCV) or anti-human immunodeficiency virus (HIV).
10. Known or suspected hypersensitivity to KM-819, or any components of the formulation(s) used.
11. Patient has a serious medical or surgical condition.
12. Patients unable to understand the consent form, and determined by investigator with too serious problems for participating in the study.
13. Patients unable to visit the clinical site on schedule due to the no ability mobilize.
14. Patients who had brain surgery history.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2024-08-19 (Actual); Study Completion 2024-08-19 (Actual)

PRIMARY OUTCOMES:
Percentage change from baseline in putaminal [18F]FP-CIT (18F-FP-CIT Positron Emission Tomography for Correlating Motor and Cognitive Symptoms of Parkinson's Disease) binding | From Baseline to Week 36
  To evaluate the efficacy of KM-819 compared to placebo in subjects with MSA for slowing the progression of MSA. The putaminal [18F]FP-CIT binding will allow quantification of MSA progression during 36 weeks.

SECONDARY OUTCOMES:
Change from baseline in the Unified Multiple System Atrophy Rating Scale (UMSARS) scores (UMSARS I + II) | From Baseline to Week 36
  To evaluate the efficacy of KM-819 compared to placebo in subjects with MSA for slowing the progression of MSA. The Unified Multiple System Atrophy Rating Scale (UMSARS) was developed to provide a surrogate measure of disease progression in multiple system atrophy. It is composed of four subscales: UMSARS-I (12 items) rates patient-reported functional disability (Historical Review), UMSARS-II (14 items) assesses motor impairment based on a clinical examination. Each item scores 0-4. UMSARS-I total score is 48 and UMSARS-II total score is 56. Higher scores on the UMSARS indicate greater disability.
Change from baseline in the UMSARS I scores | From Baseline to Week 36
  To evaluate the efficacy of KM-819 compared to placebo in subjects with MSA for slowing the progression of MSA. The Unified Multiple System Atrophy Rating Scale (UMSARS) was developed to provide a surrogate measure of disease progression in multiple system atrophy. It is composed of four subscales: UMSARS-I (12 items) rates patient-reported functional disability (Historical Review), UMSARS-II (14 items) assesses motor impairment based on a clinical examination. Each item scores 0-4. UMSARS-I total score is 48. Higher scores on the UMSARS indicate greater disability.
Change from baseline in the UMSARS II scores | From Baseline to Week 36
  To evaluate the efficacy of KM-819 compared to placebo in subjects with MSA for slowing the progression of MSA. The Unified Multiple System Atrophy Rating Scale (UMSARS) was developed to provide a surrogate measure of disease progression in multiple system atrophy. It is composed of four subscales: UMSARS-I (12 items) rates patient-reported functional disability (Historical Review), UMSARS-II (14 items) assesses motor impairment based on a clinical examination. Each item scores 0-4. UMSARS-II total score is 56. Higher scores on the UMSARS indicate greater disability.
Percentage change from baseline in putaminal glucose metabolism | From Baseline to Week 36
  To evaluate the efficacy of KM-819 compared to placebo for slowing the putaminal of MSA, as measured by [18F]FDG PET (fluorodeoxyglucose (FDG)-positron emission tomography (PET)).
Percentage change from baseline in cerebellar glucose metabolism | From Baseline to Week 36
  To further evaluate the efficacy of KM-819 compared to placebo for slowing the cerebellar progression of MSA, as measured by [18F]FDG PET.
Change from baseline in the Unified Parkinson Disease Rating Scale (UPDRS) III score | From Baseline to Week 36
  To evaluate the efficacy of KM-819 compared to placebo in subjects with MSA for slowing the progression of MSA, measured by clinical scales. The UPDRS is the most widely applied rating instrument for PD. The Total UPDRS III scale includes 18 items. Each item scores 0-4. UPDRS III total score is 72. The highest score refers to the most severe level of disability due to Parkinson's disease.
Change from baseline in the Scale for the Assessment and Rating of Ataxia (SARA) score | From Baseline to Week 36
  To evaluate the efficacy of KM-819 compared to placebo in subjects with MSA for slowing the progression of MSA, measured by clinical scales. The SARA is a tool for assessing ataxia. It has eight categories with an accumulative scores ranging from 0 (no ataxia) to 40 (most severe ataxia). The eight categories were: Gait (0-8 score); Stance (0-6 score); Sitting (0-4 score); Speech disturbance (0-6 score); Finger chase(0-4 score); Nose-finger test (0-4 score); Fast alternating hand movements (0-4 score); Heel-shin slide (0-4 score). Mild dependence: 5.5 or lower, Moderate dependence: 14.25 or lower, Maximal dependence: 23 of higher.
Change from baseline in the Montreal Cognitive Assessment (MoCA) score | From Baseline to Week 36
  To evaluate the efficacy of KM-819 compared to placebo in subjects with MSA for slowing the progression of MSA, measured by clinical scales. MoCA can be used to detect dementia in a clinical setting. A total score of 30 with over 26 is normal. The lower score refers the severe cognitive impairment.
Change from baseline in the Beck's Depression Inventory (BDI-II) score | From Baseline to Week 36
  To evaluate the efficacy of KM-819 compared to placebo in subjects with MSA for slowing the progression of MSA, measured by clinical scales. The BDI-II is scored by summing the ratings for the 21 items. Each item is rated on a 4-point scale ranging from 0 to 3. The maximum total score is 63. Measures of 0-13: Minimal, 14-19: Mild, 20-28: Moderate, 29-63: Severe.
Number of subjects with adverse events (AEs) and serious AEs (SAEs) | From Screening (Day -4) to Week 40
  To evaluate the safety of KM-819 in subjects with MSA.
Maximum observed concentration (Cmax) | From Baseline to Week 36
  To describe the pharmacokinetics parameter (Cmax) of KM-819 using sparse PK sampling.
Area under the concentration-time curve (AUC) | From Baseline to Week 36
  To describe the pharmacokinetics parameter (AUC) of KM-819 using sparse PK sampling.
Time of maximum observed concentration (Tmax) | From Baseline to Week 36
  To describe the pharmacokinetics parameter (Tmax) of KM-819 using sparse PK sampling.

CONTACTS AND LOCATIONS:
Overall Officials: Chong Sik Lee, Principal Investigator — PI
Locations (1):
- CHA Bundang Medical Center, CHA University, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided